CLINICAL TRIAL: NCT03903783
Title: Impact of Cefotaxime and Ceftriaxone on the Emergence and Carrying of Multidrug-Resistant Bacteria and Relationship to Residual Antibiotic Levels in Stool
Brief Title: Impact of Cefotaxime and Ceftriaxone on the Emergence and Carrying of Multidrug-Resistant Bacteria
Acronym: CROCTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CROCTX
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections | interventions — Cefotaxime; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefotaxime (Active Comparator)
  Interventions: Other: Cefotaxime
- Ceftriaxone (Active Comparator)
  Interventions: Other: Ceftriaxone

INTERVENTIONS:
Other: Cefotaxime — Patients with C3G antibiotic therapy will receive cefotaxime. On the day of inclusion (T0, + 24 hours), a stool culture is performed on the first stool issued after the start of antibiotic therapy to detect BMR carriage and to evaluate the initial flora and fecal abundance initial relative in culturable multiresistant bacteria. In the absence of stool emission by the patient, an eswab rectal swab will be performed.
  72 hours (± 24 hours, T1) after the start of antibiotic therapy, a stool sample will be taken and at the end of antibiotic therapy (+ 24 hours, T2) or during the oral relay to evaluate the modification of the initial flora and the relative fecal abundance of culturable multiresistant bacteria. In the case of "normal" transit (daily bowel movement), the bowel movement 72 hours after the start of antibiotic therapy will be analyzed. In the absence of stool emission by the patient, an eswab rectal swab will be performed.
  Arms: Cefotaxime
Other: Ceftriaxone — Patients with C3G antibiotic therapy will receive ceftriaxone. On the day of inclusion (T0, + 24 hours), a stool culture is performed on the first stool issued after the start of antibiotic therapy to detect BMR carriage and to evaluate the initial flora and fecal abundance initial relative in culturable multiresistant bacteria. In the absence of stool emission by the patient, an eswab rectal swab will be performed.
  72 hours (± 24 hours, T1) after the start of antibiotic therapy, a stool sample will be taken and at the end of antibiotic therapy (+ 24 hours, T2) or during the oral relay to evaluate the modification of the initial flora and the relative fecal abundance of culturable multiresistant bacteria. In the case of "normal" transit (daily bowel movement), the bowel movement 72 hours after the start of antibiotic therapy will be analyzed. In the absence of stool emission by the patient, an eswab rectal swab will be performed.
  Arms: Ceftriaxone

SUMMARY:
Among enterobacteria, the production of ESBL is the first cause of multidrug resistance. The first cases of ESBL-producing enterobacteriaceae (EBLSE) infections were described during the 1980s and subsequently experienced global spread. Since the beginning of the century, the prevalence of EBLSE infections, especially among E. coli and K. pneumoniae, has increased dramatically. The emergence of multidrug-resistant enterobacteria is currently posing a real public health problem. The European antimicrobial resistance surveillance network evaluated, among clinical strains, the resistance rate for 3rd generation cephalosporins (C3G) at 9.5% for Escherichia coli and 28% for Klebsiella pneumoniae. The consequences of multidrug-resistant enterobacterial infections, which are mainly represented by ESBLs, are currently well known, both from the individual point of view (increase in mortality and length of hospital stay) and collective (increase of costs of care).

Data from the literature reveal an increased risk of ESBL bacteremia in patients with rectal carriage of ESBL-producing enterobacteria. The study by Goulenok et al. found as a risk factor for EBLSE bacteremia in patients known to be carriers at the rectal level the existence of antibiotic selection pressure and the presence of a urinary catheter. Woerther et al. have explained in their work that the digestive microbiota confers resistance to colonization by BMR. The impact of antibiotics on the latter leads to a probable rupture of this barrier and a loss of this resistance to colonization. In addition, each antibiotherapy does not impact the digestive microbiota equally and it seems that antibiotics with high anti-anaerobic activity or high biliary elimination are the most impacting. It is therefore essential, at a time of multidrug resistance, to focus on the influence of antibiotics on the digestive microbiota and the emergence and carriage of BMR.

Ceftriaxone and cefotaxime are two injectable injectable third-generation cephalosporins (C3G) commonly used in clinical practice. Despite their similar spectrum of action, it should be noted that they have substantially different pharmacokinetic properties, especially with regard to their half-life and their elimination routes (mainly urinary for cefotaxime, mixed: biliary and urinary for ceftriaxone). Some works have already been interested in this topic. Grohs et al. carried out a comparative study between ceftriaxone and cefotaxime on the emergence of AmpC hyperproducing enterobacteria (HL-CASE). This single-site study demonstrated that, at a hospital level, the preferential use of cefotaxime rather than ceftriaxone had collective and ecological benefits at the service level. Indeed, their results conclude that resistance development is weaker, as well as more limited carriage of HL-CASE Enterobacterial strains by replacing ceftriaxone with cefotaxime. It should be noted, however, that the modification of prescribing practices of C3G has been coupled with various measures to limit the emergence of AmpC hyperproductive enterobacteria (reinforcement of hygiene rules, awareness of the health care team at EBLSE, control of antibiotic ...).

In a context where the emergence of multidrug-resistant bacteria continues to increase, it seems appropriate to conduct a study to compare the impact of the use of ceftriaxone or cefotaxime on the emergence of BMR at the individual level. In the absence of a study clearly establishing the link between C3G types (ceftriaxone, cefotaxime) and the emergence of BMR and in line with the above research, this study aims to compare the microbiological impact of the use of either of these two C3Gs (in terms of emergence of bacterial resistance and impact on the diversity and quantity of digestive digestive bacteria). The study will have two periods: Period 1 during which patients hospitalized in the emergency department or in internal medicine and receiving C3G antibiotics will receive ceftriaxone, and the period 2 during which cefotaxime is cephalosporin used in first intention in these same patients.

Thus, this research project, by focusing on these 5 parameters in patients treated with ceftriaxone or cefotaxime, should make it possible to prove the influence of these antibiotherapies on the carriage of BMR (deleterious action on the diversity and the quantity of the intestinal bacterial flora, resulting in an increase in the relative fecal abundance of these BMRs promoting their carriage). In addition, the hypothesis is that, contrary to current data, cefotaxime is found at sufficiently high concentrations in the feces to have an impact on the microbiota equivalent to that of ceftriaxone, despite less significant biliary elimination.

This study therefore aims to compare their impacts on the microbiota and in particular on the emergence of multidrug-resistant bacteria (BMR) and enteropathogens such as Clostridium difficile.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient hospitalized in the department of internal medicine within the Hospital Group Paris Saint-Joseph
* Patient with probabilistic or documented C3G infection
* Patient affiliated to a social security scheme
* Francophone patient
* Patient living at home, in a nursing home or retirement home
* Patient able to give free, informed and express consent

Exclusion Criteria:

* Patient with allergy to cephalosporins
* Inclusion time greater than 24 hours after initiation of antibiotic therapy
* Patient having been hospitalized in the 3 months preceding the inclusion
* Patient who received antibiotic treatment within 3 weeks prior to inclusion
* Patient being included in another study
* Pregnant woman
* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Emergence of enterococci resistant to vancomycin | 24 Hours after the end of atnibiotherapy
Emergence of EBLSE | 24 Hours after the end of atnibiotherapy
Emergence of Clostridium difficile | 24 Hours after the end of atnibiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France